CLINICAL TRIAL: NCT04912310
Title: Efficacy Evaluation and Influencing Factors of Argon Laser Peripheral Iridoplasty in Acute Angle Closure Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-480
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-07

CONDITIONS: Acute Angle-Closure Glaucoma
Keywords: Acute angle-closure glaucoma; Argon laser peripheral iridoplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute angle closure glaucoma (Experimental): Argon laser peripheral iridoplasty
  Interventions: Device: Argon laser peripheral iridoplasty

INTERVENTIONS:
Device: Argon laser peripheral iridoplasty — Argon laser peripheral iridoplasty was performed in patients with severe acute angle closure glaucoma whose intraocular pressure could not be controlled by medication

SUMMARY:
To investigate the changes of angle structure and intraocular pressure after argon laser peripheral iridoplasty in patients with acute angle closure glaucoma patients whose intraocular pressure could not be controlled by drug therapy during the major attack period.

DETAILED DESCRIPTION:
To evaluate intraocular pressure and anterior segment optical coherence tomography measurement parameters at baseline and each follow-up. Each patient was followed up for 6 weeks for 9 times. Visit 1st was baseline examination, visit 2nd was 1 hour after argon laser peripheral iridoplasty treatment, visit 3rd was 2 hours after argon laser peripheral iridoplasty treatment, visit 4th was 1 week after argon laser peripheral iridoplasty treatment, visit 5th was 2 week after argon laser peripheral iridoplasty treatment, and visit 6th was 1 month after argon laser peripheral iridoplasty treatment, visit 7th was 6 week after argon laser peripheral iridoplasty treatment.

ELIGIBILITY:
Inclusion Criteria:

* One eye had an acute attack, which could not be relieved by medication, and the intraocular pressure was more than 21mmhg;
* The patients were 40 to 80 years old, regardless of gender;
* Patients are able and willing to comply with the research guidance and may complete all visits required by the research;
* Informed consent has been signed.

Exclusion Criteria:

* History of ocular trauma;
* Any previous intraocular surgery;
* Secondary glaucoma was diagnosed, including uveitis, neovascular glaucoma, glaucoma with elevated superior scleral venous pressure, lens dissolution glaucoma, glaucoma caused by lens dislocation, lens cortical glaucoma, pigmented glaucoma, etc;
* The patient's history indicated that he had severe dysfunction of heart, lung, liver and kidney;
* Women in pregnancy, lactation or planned pregnancy;
* The researchers believe that the patient's condition may put the patient at a significant risk, may confuse the results of the study, or may significantly interfere with the patient's participation in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 6 weeks
  Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: kaijun wang, MD, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Eye center, 2nd Affiliated Hospital, School of Medicine, Zhejiang University,, Hangzhou, Zhejiang, China